CLINICAL TRIAL: NCT01933139
Title: Informed Consent for Hysterectomy: Effectiveness of Audio-visual Presentations on Patient Comprehension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alicia Pallett, Principal Investigator, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: ICHyst
Record Dates: First submitted 2013-08-26; First posted 2013-09-02 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Hysterectomy; Informed Consent
Keywords: Informed consent; preoperative counseling; hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Audio-visual presentation (Experimental): The intervention group will watch a 10-minute scripted video explaining the procedure, risks, benefits, expectations, and long term complications that relate to hysterectomies before face-to-face interaction with the surgeon. Patients in both arms will then sign the same standard pre-surgical informed consent form before undergoing the procedure.
  Interventions: Other: Audio-visual presentation
- Control (No Intervention): standard physician interaction (control arm)

INTERVENTIONS:
Other: Audio-visual presentation
  Arms: Audio-visual presentation

SUMMARY:
To determine whether the addition of audio-visual presentations to standard physician interaction improves patient comprehension as it relates to the information provided during the informed consent process in patients undergoing hysterectomy.

DETAILED DESCRIPTION:
Aim: To determine whether the addition of audio-visual presentations to standard physician interaction improves patient comprehension as it relates to the information provided during the informed consent process in patients undergoing hysterectomy.

Design: This is a randomized controlled trial comparing standard physician interaction (control arm) to standard physician interaction plus audio-visual presentation (experimental arm) during the informed consent process for patients undergoing hysterectomy to determine the effectiveness of audio-visual presentations on patient comprehension. All subjects will undergo knowledge questionnaires at four separate time points - prior to their preoperative appointment, immediately after their preoperative appointment, day of surgery, and at the six-week follow-up visit. The control group will be consented in the standard fashion with face-to-face interaction with their surgeon. The intervention group will watch a 10-minute scripted video explaining the procedure, risks, benefits, expectations, and long term complications that relate to hysterectomies before face-to-face interaction with the surgeon. Patients in both arms will then sign the same standard pre-surgical informed consent form before undergoing the procedure. All interactions with the physicians (control and experimental) will be audiotaped to assess the number of patient questions, the time spent with each patient, and the quality of subject material discussed in the control group. Subjects will also receive satisfaction questionnaires after the preoperative visit.

Setting: Research will take place in the gynecology clinic and surgical suites of San Antonio Military Medical Center.

Subjects: Approximately 120 subjects will be recruited from the San Antonio Military Medical Center gynecology clinic (50 in each arm). Eligible subjects include all patients scheduled for hysterectomy with or without salpingo-oophorectomy for benign indications, civilian and military, female only, older than 18yo, English-speaking, with intact hearing and vision, and able to provide consent without representation.

Measures: In this study, patient literacy will be determined using the REALM score (Rapid Estimate of Adult Literacy in Medicine). Patient knowledge questionnaires were created by the investigators of the study. Satisfaction will be measured by a validated questionnaire (CSQ-8). Primary objectives will be addressed through analysis of subjects' difference scores on comprehension assessments at each of four time points. Secondary objectives including patient satisfaction, time spent by physician in face-to-face interaction, questions asked by the patients, and quality of physician counseling (inclusion of key items in control arm) will also be analyzed between groups.

ELIGIBILITY:
Inclusion Criteria:

* All adult female patients undergoing vaginal, abdominal, or laparoscopic hysterectomy with or without salpingo-oophorectomy for benign indications

Exclusion Criteria:

* malignant indication for the surgery
* vision- and/or hearing-impairment
* unwilling or unable to provide consent
* under age 18
* not primarily English-speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Patient comprehension | 6 weeks
  the effectiveness of an audio-visual presentation in conjunction with the standard physician-patient interaction on patient comprehension as it pertains to the informed consent process prior to undergoing hysterectomy

SECONDARY OUTCOMES:
Patient satisfaction | 1 day
  Satisfaction will be measured by a validated questionnaire (CSQ-8) to determine whether higher patient satisfaction in experimental (audio-visual) arm.
Physician efficiency | 1 day
  Doctor-patient interactions will be timed for all subjects by extrapolating from audiotaped encounters.
Adequacy and quality of the physician-directed informed consent process | 1 day
  Physicians giving informed consent without the audio-visual intervention will be assessed through audiotaping of their discussion to see if discussion includes standardized preoperative checklist items.

CONTACTS AND LOCATIONS:
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States